CLINICAL TRIAL: NCT03272620
Title: Atrial Fibrillation Registry at the Emergency Department of the Medical University of Vienna: A Tool for Structured Diagnosis and Treatment
Brief Title: Atrial Fibrillation at the Viennese University Emergency Department
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexander Spiel, Associate Professor at the Department of Emergency Medicine, Medical University of Vienna
Other Study IDs: 98765
Record Dates: First submitted 2017-08-23; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The results of this study could imply that a atrial fibrillation registry, as a tool for structured diagnosis and therapy in patients with atrial fibrillation, may improve patient care for this rapidly growing population.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common cardiac arrhythmia and is associated with increased cardiovascular morbidity and mortality, with stroke being an especially important and potentially devastating complication. The number of patients with atrial fibrillation is likely to increase 2.5-fold during the next 50 years, reflecting the growing proportion of elderly individuals. Emergency departments play a central role in diagnosis and treatment (rhythm and rate control, initiation of anticoagulatory therapy for stroke prevention) of atrial fibrillation. Additionally, embolic (e.g. stroke, mesenteric ischemia) complications of atrial fibrillation and bleeding complications (e.g. gastrointestinal and intracranial) of anticoagulatory therapy are likewise treated at emergency departments.

Therefor the investigators hypothesis implies that the atrial fibrillation registry could serve as a tool for structured diagnosis and therapy in patients with atrial fibrillation and therefore may improve patient care. Additionally, diagnostic and therapeutic shortcomings by analyzing registry data may be detected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation treated at the Emergency Department of the Medical University of Vienna
* Signed consent

Exclusion Criteria:

* Inclusion criteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation treated at the Emergency Department of the Vienna Medical University. Currently, about 600 patients with atrial fibrillation are seen annually at the Emergency Department, every patient with atrial fibrillation treated at the Emergency Department should be included.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-10-22 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major adverse cardiac events | Follow up (10 years)
  frequency distribution

SECONDARY OUTCOMES:
Number of successfully conducted cardioversions | Follow up (10 years)
  frequency distribution

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Spiel, Priv. Doz., Principal Investigator — Medical University Vienna
Locations (1):
- Emergency Department, Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Risk factors for stroke and efficacy of antithrombotic therapy in atrial fibrillation. Analysis of pooled data from five randomized controlled trials. Arch Intern Med. 1994 Jul 11;154(13):1449-57. PMID 8018000
- [Background] Lip GY, Tean KN, Dunn FG. Treatment of atrial fibrillation in a district general hospital. Br Heart J. 1994 Jan;71(1):92-5. doi: 10.1136/hrt.71.1.92. PMID 8297706
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] O'Reilly DJ, Hopkins RB, Healey JS, Dorian P, Sauriol L, Tarride JE, Burke N, Goeree RA. The burden of atrial fibrillation on the hospital sector in Canada. Can J Cardiol. 2013 Feb;29(2):229-35. doi: 10.1016/j.cjca.2012.03.023. Epub 2012 May 30. PMID 22652091
- [Background] Domanovits H, Schillinger M, Thoennissen J, Nikfardjam M, Janata K, Brunner M, Laggner AN. Termination of recent-onset atrial fibrillation/flutter in the emergency department: a sequential approach with intravenous ibutilide and external electrical cardioversion. Resuscitation. 2000 Aug 1;45(3):181-7. doi: 10.1016/s0300-9572(00)00180-5. PMID 10959017
- [Background] Vinson DR, Hoehn T, Graber DJ, Williams TM. Managing emergency department patients with recent-onset atrial fibrillation. J Emerg Med. 2012 Feb;42(2):139-48. doi: 10.1016/j.jemermed.2010.05.017. Epub 2010 Jul 15. PMID 20634022
- [Background] von Besser K, Mills AM. Is discharge to home after emergency department cardioversion safe for the treatment of recent-onset atrial fibrillation? Ann Emerg Med. 2011 Dec;58(6):517-20. doi: 10.1016/j.annemergmed.2011.06.014. Epub 2011 Jul 29. PMID 22098994
- [Background] Bellone A, Etteri M, Vettorello M, Bonetti C, Clerici D, Gini G, Maino C, Mariani M, Natalizi A, Nessi I, Rampoldi A, Colombo L. Cardioversion of acute atrial fibrillation in the emergency department: a prospective randomised trial. Emerg Med J. 2012 Mar;29(3):188-91. doi: 10.1136/emj.2010.109702. Epub 2011 Mar 21. PMID 21422032
- [Background] Hochtl T, Huber K. New anticoagulants for the prevention of stroke in atrial fibrillation. Fundam Clin Pharmacol. 2012 Feb;26(1):47-53. doi: 10.1111/j.1472-8206.2011.00982.x. Epub 2011 Aug 29. PMID 21883447
- [Background] Oldgren J, Healey JS, Ezekowitz M, Commerford P, Avezum A, Pais P, Zhu J, Jansky P, Sigamani A, Morillo CA, Liu L, Damasceno A, Grinvalds A, Nakamya J, Reilly PA, Keltai K, Van Gelder IC, Yusufali AH, Watanabe E, Wallentin L, Connolly SJ, Yusuf S; RE-LY Atrial Fibrillation Registry Investigators. Variations in cause and management of atrial fibrillation in a prospective registry of 15,400 emergency department patients in 46 countries: the RE-LY Atrial Fibrillation Registry. Circulation. 2014 Apr 15;129(15):1568-76. doi: 10.1161/CIRCULATIONAHA.113.005451. Epub 2014 Jan 24. PMID 24463370
- [Background] Rovellini A, Folli C, Cardani F, Monzani V. Thromboembolic and haemorrhagic events in permanent atrial fibrillation: observational study in an emergency department. Eur J Intern Med. 2009 Dec;20(8):756-9. doi: 10.1016/j.ejim.2009.08.008. Epub 2009 Sep 24. PMID 19892303
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines-CPG; Document Reviewers. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation--developed with the special contribution of the European Heart Rhythm Association. Europace. 2012 Oct;14(10):1385-413. doi: 10.1093/europace/eus305. Epub 2012 Aug 24. No abstract available. PMID 22923145
- [Derived] Niederdockl JD, Simon A, Buchtele N, Schutz N, Cacioppo F, Oppenauer J, Gupta S, Lutnik M, Schnaubelt S, Spiel A, Roth D, Wimbauer F, Fegers-Wustrow I, Esefeld K, Halle M, Scharhag J, Laschitz T, Herkner H, Domanovits H, Schwameis M. Prediction of Successful Pharmacological Cardioversion in Acute Symptomatic Atrial Fibrillation: The Successful Intravenous Cardioversion for Atrial Fibrillation (SIC-AF) Score. J Pers Med. 2022 Mar 30;12(4):544. doi: 10.3390/jpm12040544. PMID 35455660
- [Derived] Niederdockl J, Simon A, Cacioppo F, Buchtele N, Merrelaar A, Schutz N, Schnaubelt S, Spiel AO, Roth D, Schorgenhofer C, Herkner H, Domanovits H, Schwameis M. Predicting spontaneous conversion to sinus rhythm in symptomatic atrial fibrillation: The ReSinus score. Eur J Intern Med. 2021 Jan;83:45-53. doi: 10.1016/j.ejim.2020.07.022. Epub 2020 Sep 18. PMID 32951957
- [Derived] Niederdockl J, Simon A, Schnaubelt S, Schuetz N, Laggner R, Sulzgruber P, Spiel AO, Herkner H, Laggner AN, Domanovits H. Cardiac biomarkers predict mortality in emergency patients presenting with atrial fibrillation. Heart. 2019 Mar;105(6):482-488. doi: 10.1136/heartjnl-2018-313145. Epub 2018 Nov 10. PMID 30415208